CLINICAL TRIAL: NCT02354612
Title: An Open Label Continuation Study of TRC105 Therapy for Patients Who Have Completed a Prior TRC105 Trial and Are Judged by the Investigator to Have the Potential to Benefit From Continued TRC105 Therapy
Brief Title: Open Label Continuation Study of TRC105 for Patients Who Have Completed a Prior TRC105 Trial
Status: No longer available | Type: Expanded Access
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 105CON101
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — carotuximab; Bevacizumab; Axitinib; pazopanib; Capecitabine

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: TRC105
  Other Names: Chimeric Antibody (TRC105) to CD105
Drug: Bevacizumab — companion therapy selection depends on companion therapy used in the parent study
  Other Names: Avastin
Drug: Axitinib — companion therapy selection depends on companion therapy used in the parent study
  Other Names: Inlyta
Drug: Pazopanib — companion therapy selection depends on companion therapy used in the parent study
  Other Names: Votrient
Drug: Capecitabine — companion therapy selection depends on companion therapy used in the parent study
  Other Names: Xeloda

SUMMARY:
Open-label, continuation study

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-randomized, study of TRC105 in patients that have completed a previous TRC105 study and are judged by the investigator to have the potential to benefit from continued TRC105 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a TRACON Pharmaceuticals sponsored parent TRC105 study and, thought to have potential to derive clinical benefit from continued treatment with TRC105 in the opinion of the parent study investigator.
* Willing and able to consent for self to participate in study
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* 18 years of age or older
* ability to begin TRC105 dosing on this protocol within 6 weeks from the subjects last dose of TRC105 in the parent TRC105 study

Exclusion Criteria:

* Any clinical event that would make TRC105 therapy inappropriate under the parent protocol
* Current treatment in another clinical study
* Pregnant or breastfeeding
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator, would make the subject inappropriate for entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD, Study Director — Tracon Pharmaceuticals Inc.
Locations (1):
- UCLA, Santa Monica, California, United States